CLINICAL TRIAL: NCT00267631
Title: The Influence of Childhood Obesity on Presentation to a Pediatric Emergency Department
Brief Title: Impact of Body Weight on the Immediate Health of the Pediatric Population
Status: Completed | Type: Observational
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 05-02-VA10
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-07

CONDITIONS: Childhood Obesity
Keywords: children, obesity, emergency medicine
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- At Risk Body Weight: Children with a BMI greater and equal to 85%
- Normal Body Weight: Children with a BMI of 25 to 75%

SUMMARY:
Objective: Obesity amongst children is a public health issue in the United States and is rising at an alarming rate. The purpose of this study is to determine if there is any correlation between At Risk body weight (overweight and obese) and immediate health of the pediatric population.

Methodology: As part of routine patient care, we measured length in addition to weight of patients 2 years to 18 years of age presenting to the pediatric emergency department. A report was run monthly to calculate the BMI of all patients for whom data is available. The data were plotted on the year 2000 gender based BMI for age percentile growth charts from CDC. A retrospective electronic chart review was conducted for patients At Risk body weight (BMI ≥ 85%), and were compared to "control" or healthy (BMI of 25 - 75 %) group for six groups of final ED diagnoses of infectious diseases.

DETAILED DESCRIPTION:
A. Background and Significance:

Obesity is a public health issue in the United States. Obesity amongst children is rising at an alarming rate. Thirty percent of US children aged 6 to 19 are over weight and 15 % are obese1. It is estimated that over 18 million US children are over weight. The long-term impact of childhood obesity on such diseases as Diabetes, Asthmaand Hypertension, is well studied. The effects of childhood obesity on the current health status of the pediatric population have not been studied.

B. Methodology:

As part of routine patient care, we measured length in addition to weight of patients 2 years to 18 years of age presenting to the pediatric emergency department. A report was run monthly to calculate the BMI of all patients for whom data is available. The data were plotted on the year 2000 gender based BMI for age percentile growth charts from CDC. A retrospective electronic chart review was conducted for patients At Risk body weight (BMI ≥ 85%), and were compared to "control" or healthy (BMI of 25 - 75 %) group for six groups of final ED diagnoses of infectious disease (ID). Data were entered and analyzed via SPSS 14.0 for Windows 2000 software systems.

ELIGIBILITY:
Inclusion Criteria:Age 2-18 yrs for whom a length and weight is possible -

Exclusion Criteria:Under 2 yrs or over 18 yrs of age or inability to weigh and measure pt

-

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric Emergency Medicine Patients
Sampling Method: Non-Probability Sample
Enrollment: 5392 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estevan Garcia, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric Emergency Department
Pre-assignment Details: No significant events
Groups:
- At Risk Body Weight: Children with BMI greater and equal to 85%
- NOrmal Body Weight: Children with BMI of 25-75%
Period: Overall Study
Arm/Group | At Risk Body Weight | NOrmal Body Weight
Started | 2361 | 3031
Completed | 2361 | 3031
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- At Risk Body Weight: Children with BMI greater adn equal to 85%
- Total: Total of all reporting groups
Arm/Group | At Risk Body Weight | Normal Body Weight | Total
Number analyzed (Participants) | 3031 | 2361 | 5392
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3031 | 2361 | 5392
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.2 (4.3) | 8.8 (4.7) | 9.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1229 | 1031 | 2260
  Male | 1802 | 1330 | 3132
Region of Enrollment [Number; unit: participants]
  United States | 3031 | 2361 | 5392

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis of Infectious Disease
Description: The Children visiting the ED having an infectious disease
Time Frame: 30 minutes
Measure: Number; unit: Participants
Arm/Group | At Risk Body Weight | Normal Body Weight
Number analyzed (Participants) | 2361 | 3031
Participants | 900 | 1067
Statistical Analysis 1: Comparison: At Risk Body Weight vs Normal Body Weight; Test type: Superiority or Other; p = .026, Chi-squared

ADVERSE EVENTS:
Arm/Group | At Risk Body Weight | Normal Body Weight
Serious Adverse Events (participants affected / at risk) | 0/3031 | 0/2361
Other Adverse Events (participants affected / at risk) | 0/3031 | 0/2361

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No